Cognitive Training with and without tDCS to Improve Cognition in HIV

December 2, 2014

Statistical Analysis Plan

Study outcomes will be evaluated through analysis of group differences on neuropsychological measures after correction for baseline differences in age, disease status (CD4 count), mood, and baseline performance. Additional outcomes will include the rate of learning in the computer-delivered memory and attention task between groups. Individual and group slopes for the task will be plotted and visually inspected as well as tested using parametric statistics.